CLINICAL TRIAL: NCT03840083
Title: What is Sleep's Role in Alzheimer's Disease? Insight From Healthy Aging
Brief Title: Sleep-dependent Learning in Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Rebecca Spencer, Professor, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-4290
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Sleep
MeSH Terms: interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep (Experimental): Individuals will either nap (Exps 1, 4) or have overnight sleep (Exps 2, 3, 5, 6)
  Interventions: Behavioral: Sleep
- Wake (No Intervention): Individuals will stay awake for the same amount of time as they slept in the sleep condition

INTERVENTIONS:
Behavioral: Sleep — Participants will sleep (either a mid-day nap or normal overnight sleep)
  Arms: Sleep

SUMMARY:
The specific objective of this proposed research is to understand whether deficits in sleep-dependent memory changes reflect age-related changes in sleep, memory, or both. The central hypothesis is that changes in both memory and sleep contribute to age-related changes in sleep-dependent memory processing. To this end, the investigators will investigate changes in learning following intervals of sleep (overnight and nap) and wake in young and older adults.

DETAILED DESCRIPTION:
Exp 1: Using neuroimaging, the investigators will consider whether differences in brain areas engaged during memory encoding contribute to age-related changes in sleep-dependent memory consolidation for a word-pair learning task.

Exp 2: The investigators will examine the rate of memory decay between encoding and sleep using two probes of declarative memory (word-pair learning and visuo-spatial learning).

Exp 3: The investigators will provide additional opportunity for encoding of the word-pair and visuo-spatial learning tasks.

Exp 4: Using neuroimaging, the investigators will examine neural engagement during encoding and performance following intervals of sleep and wake.

Exp 5: The investigators will examine the rate of decay of motor sequence learning.

Exp 6: The investigators will examine whether enhanced training ('overtraining') improves sleep-dependent memory consolidation for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 yrs
* Healthy sleeper
* No diagnosed sleep or neurodegenerative disorder

Exclusion Criteria:

1. Past diagnosis of any sleep disorder or evidence of a sleep disorder as assessed by self-reported sleep quality assessments, a standardized diagnostic interview, and an acclimation night of polysomnography. Using acclimation-night polysomnography, participants will be excluded with an Apnea-Hypopnea Index >15; a Period-Limb Movement in Sleep index of >15/hr; sleep-onset latency > 45 min (indicative of insomnia); or sleep efficiency < 80% (see Edinger et al., Sleep, 2004). In cases in which questions arise regarding a participants' inclusion or sleep records, a practicing neurologist board-certified in sleep medicine will review the documentation.
2. Past diagnosis neurological illness or head injury
3. Reported average sleep per night < 5 or > 9 hrs
4. Current employment involving shift work or an inability to keep a regular sleep schedule during the week prior to testing
5. Current use of psychotropic, recreational drugs, or sleep-altering medications (sleep medications, cold medicines within the past week, clonidine, sympathomimetic stimulants)
6. Daily caffeine intake of > 4 cups (coffee, tea, colas)
7. Weekly alcohol intake of > 10 cups
8. Pregnancy or < 12 months post-partum
9. History of bipolar disorder, mania, or current evidence of depression as measured by Beck Depression Inventory score > 25
10. Abnormal sleep (e.g., shift work, travel across >2 time zones within the past 3 months).
11. Diagnosis of any Axis I disorder, neurological illness or head injury (according to Demographic and Health History form);
12. Score indicative of cognitive dysfunction (subtest scores < 40)
13. Beck Depression Scale score indicative of depression (> 19).

Additionally, individuals will be excluded from magnetic resonance imaging studies (Exps 1, 4) for:

1. Left handed or ambidextrous
2. Claustrophobia
3. Presence of metal (thoroughly screened via questionnaire and metal detector)
4. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in memory accuracy for intervention compared to control | 2 hours (Experiments 1,4) or 12 hours (Experiments 2,3,5,6)
  We will measure memory accuracy before the sleep/wake interval and subtract this from memory accuracy after the sleep wake interval. If sleep benefits memory then this value will be greater in the sleep condition compared to the wake condition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No